CLINICAL TRIAL: NCT05976191
Title: Istanbul University Cerrahpaşa-IUC
Brief Title: Comparison of Fasting Blood Glucose Measurements From Fingertip and Intravenous on Patient Satisfaction in Patients With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, AYSEGUL, principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/476
Record Dates: First submitted 2023-07-20; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Fear of finger piercing; patient satisfaction; blood glucose measurement
MeSH Terms: conditions — Diabetes Mellitus; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Crossover Assignment This research was designed in a pretest posttest randomized controlled experimental type
Who Masked: Participant
Masking Description: Single (Participant) Identity information of the patients was concealed and verbal and written consents were obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients whose blood glucose is measured intravenously and from the fingertip
  Interventions: Behavioral: Patients whose blood glucose is measured intravenously and from the fingertip
- control group (No Intervention): Patients with fingertip blood glucose measurement

INTERVENTIONS:
Behavioral: Patients whose blood glucose is measured intravenously and from the fingertip — A satisfaction survey will be conducted after these patients have previously examined their blood glucose via intravenous route, then fingertip blood glucose will be measured and a satisfaction survey will be applied.
  Arms: experimental group

SUMMARY:
The study was designed as a randomized controlled experimental study in order to compare the fasting blood glucose values measured by puncturing the fingertips and using the intravenous route of patients diagnosed with diabetes mellitus, and to determine the effect on patient satisfaction. The blood glucose measurement via the intravenous catheter has an effect on increasing the comfort of the patient compared to the fingertip measurement. It is thought that information can be provided to increase patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* No advanced hearing and vision problems
* Able to speak and understand Turkish
* Easy to communicate
* literate
* Agreeing to participate in the research voluntarily
* Patients who are hospitalized
* Regular finger blood sugar monitoring,
* Patients with an intravenous vascular access date within the first 24 hours
* Patients who had been diagnosed with Type 2 Diabetes Mellitus for at least one year were.

Exclusion Criteria:

* Those who are treated with sedative drugs
* Patients using antipsychotic medication
* Patients with continuous drug infusion through the intravenous line
* Patients whose intravenous vascular access date has passed 24 hours
* Patients in unconscious, confused, apathetic state

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Measurement Patient Satisfaction Form | four months
  Does intravenous blood glucose measurement have a positive effect on patient satisfaction compared to fingertip blood glucose measurement?

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa (IUC), Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No